CLINICAL TRIAL: NCT06223386
Title: Total Lifestyle Reconstruction for Body Weight Control and Maintenance: an On-line Randomized Controlled Trial
Brief Title: Total Lifestyle Reconstruction for Body Weight Control and Maintenance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academia Sinica, Taiwan (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Wen-Harn Pan, Distinguished Research Fellow, Academia Sinica, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AS-IRB-BM-23059; EC1121001-E (Other: NHRI IRB)
Record Dates: First submitted 2024-01-12; First posted 2024-01-25 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Referral and Consultation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Traditional model (Placebo Comparator): Designed course A with 3-month consultation with the dietitians
  Interventions: Behavioral: Designed on-line course A with 3-month consultation with the dietitian
- Multi-oriented lifestyle education (Experimental): Designed course B with 3-month consultation with the dietitians
  Interventions: Behavioral: Designed on-line course B with 3-month consultation with the dietitian
- Multi-oriented lifestyle education with dietary assessment (Experimental): Designed course B with 3-month consultation with the dietitians + 3-month daily dietary assessment by the dietitians
  Interventions: Behavioral: Designed on-line course B with 3-month consultation with the dietitians + 3-month daily dietary assessment by the dietitians
- Multi-oriented lifestyle education with longer period of dietary assessment (Experimental): Designed course B with 6-month consultation with the dietitians + 6-month daily dietary assessment by the dietitians
  Interventions: Behavioral: Designed on-line course B with 6-month consultation with the dietitians + 6-month daily dietary assessment by the dietitians

INTERVENTIONS:
Behavioral: Designed on-line course A with 3-month consultation with the dietitian — Educational materials on weight reduction will be provided at the beginning of the 3-month intervention. Participants can consult with the dietitian via the APP on their mobile phones during the intervention period. These materials will encompass dietary and physical activity guidelines by the government in Taiwan.
  Arms: Traditional model
Behavioral: Designed on-line course B with 3-month consultation with the dietitian — Educational materials on weight reduction will be provided every weekday for 8 weeks. Participants can consult with the dietitian via the APP on their mobile phones during the 3-month intervention period. These materials will encompass various aspects such as dietary habits, physical activity, and daily routines, all designed to impart online lifestyle education.
  Arms: Multi-oriented lifestyle education
Behavioral: Designed on-line course B with 3-month consultation with the dietitians + 3-month daily dietary assessment by the dietitians — Educational materials on weight reduction will be provided every weekday for 8 weeks. Participants can consult with the dietitian via the APP on their mobile phones during the 3-month intervention period. These materials will encompass various aspects such as dietary habits, physical activity, and daily routines, all designed to impart online lifestyle education. In addition, dietitians assess participants' daily diet for 3 months.
  Arms: Multi-oriented lifestyle education with dietary assessment
Behavioral: Designed on-line course B with 6-month consultation with the dietitians + 6-month daily dietary assessment by the dietitians — Educational materials on weight reduction will be provided every weekday for 8 weeks. Participants can consult with the dietitian via the APP on their mobile phones during the 6-month intervention period. These materials will encompass various aspects such as dietary habits, physical activity, and daily routines, all designed to impart online lifestyle education. In addition, dietitians assess participants' daily diet for 6 months.
  Arms: Multi-oriented lifestyle education with longer period of dietary assessment

SUMMARY:
Obesity stands as a significant health concern of the 21st century. The prevalence of obesity is steadily rising worldwide, and Taiwan is no exception, with nearly four to five out of ten individuals facing issues of overweight or obesity. Additionally, approximately 1.5% of adults suffer from morbid obesity. Presently, lifestyle interventions focusing on body control have shown limited success in maintaining an ideal weight and body composition, and they are predominantly applied within clinical settings for managing morbidly obese patients.

In response to the transformations brought about by the 3C era in connecting with the public, an effective online intervention approach holds promising potential but still requires development and validation. This project endeavors to revolve around "cultivating a healthy lifestyle" by creating educational materials on weight reduction. These materials will encompass various aspects such as dietary habits, physical activity, and daily routines, all designed to impart online lifestyle education. To facilitate the intervention, the investigators plan to employ the application "Cofit" developed by the Cofit Healthcare Inc., targeting individuals with weight reduction needs. Furthermore, the investigators aim to collect research data for the analysis of intervention effectiveness.

Over a three to six-month intervention period, the research participants will receive multifaceted lifestyle education through the online app. Certified nutritionists, trained under the program, will interact with the participants online, guiding them to make changes in their diet, physical activity, and daily routines. The ultimate goal is to help the participants achieve effective weight reduction and maintain a healthy body weight in the long term.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 24 and 35

Exclusion Criteria:

* cancer
* hospitalization
* pregnancy
* depression
* currently taking weight loss drugs
* unwilling to give up meal replacement for weight loss
* unable to cooperate with the data collection and intervention guide of this study
* stage III kidney disease or above
* diabetes
* taking medication
* participation in previous weight loss courses of Qunjian Technology Company

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Achievement rate of healthy body weight at Month 3 and 6. | Baseline, Month 3 and 6
  The number of participants whose weight will be reduced to within the range of a personal BMI equal to 22 among all participants.
Change from baseline in fat percent at Month 3 and 6. | Baseline, Month 3 and 6
Change from baseline in diet quality at Month 3 and 6. | Baseline, Month 3 and 6
  Diet quality is estimated according to the daily intake of nutrients and the distribution of the six food groups, with a qualified food frequency questionnaire.
  The six food groups include:
  1. Whole grains and starchy vegetables
  2. Protein foods: soybeans, fish, eggs, and meat
  3. Vegetables
  4. Fruits
  5. Dairy
  6. Oils, nuts & seeds.

SECONDARY OUTCOMES:
Change from baseline in physical activity at Month 3 and 6. | Baseline, Month 3 and 6
Change from baseline in sleep quality at Month 3 and 6. | Baseline, Month 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Harn Pan, Ph.D., Principal Investigator — Institute of Biomedical Sciences, Academia Sinica
Locations (1):
- Institute of Biomedical Sciences, Academia Sinica, Taipei, Taiwan